CLINICAL TRIAL: NCT04286711
Title: Phase I / II Clinical Study of Albumin-paclitaxel Combined With Apatinib and Camrelizumab in the Second-line Treatment of Advanced Gastric Cancer
Brief Title: Clinical Study of Albumin-paclitaxel Combined With Apatinib and Camrelizumab in Advanced Gastric Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, Director of Department of Medical Oncology，The First Hospital of China Medical University, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-GC-I-002
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Advanced Gastric Cancer
Keywords: Apatinib Albumin-paclitaxel Camrelizumab Gastric cancer
MeSH Terms: interventions — apatinib; camrelizumab; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Albumin-paclitaxel Combined With Apatinib and Camrelizumab (Experimental): Albumin-paclitaxel: ivgtt, 75 or 100 or 125mg /m2, d1, d8; Apatinib: initial dose: 250mg,oral,once a day, after meal ( try to take the medicine at the same time each day); Camrelizumab：ivgtt, 200mg, given on the first day; Repeat the therapeutic schedule every 3 weeks
  Interventions: Drug: Albumin-paclitaxel, Apatinib, Camrelizumab

INTERVENTIONS:
Drug: Albumin-paclitaxel, Apatinib, Camrelizumab — Albumin-paclitaxel: ivgtt, 75 or 100 or 125mg /m2, d1, d8, Repeat the therapeutic schedule every 3 weeks; Apatinib: initial dose: 250mg,oral,once a day, after meal ( try to take the medicine at the same time each day); Camrelizumab：ivgtt, 200mg, given on the first day, Q3W;
  Other Names: Paclitaxel for injection（Albumin Bound），Apatinib Mesylate Tablets，SHR-1210

SUMMARY:
This study is to evaluate the tolerance of albumin paclitaxel combined with apatinib and Camrelizumab in the second-line treatment of advanced gastric cancer to determine the maximum tolerable dose (MTD) of the combination.

DETAILED DESCRIPTION:
This is a Single arm, open, phase I / II clinical trial. The study was divided into tolerance observation stage (dose exploration stage) and efficacy expansion stage (dose expansion stage).

This study is to evaluate the tolerance of albumin-paclitaxel combined with apatinib and Camrelizumab in the second-line treatment of advanced gastric cancer to determine the maximum tolerable dose (MTD) of the combination.

The secondary objective was to evaluate the safety and efficacy of albumin- paclitaxel in combination with apatinib and Camrelizumab in the second-line treatment of advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed gastric or gastroesophageal junction adenocarcinoma (GEJ).
2. Age: 18-70 years old, Female or Male.
3. Failure or intolerance of first-line chemotherapy which requires that the first-line chemotherapy regimen include the scheme based on platinum and / or fluorouracil drugs.
4. ECOG performance status 0-1.
5. Patients must have at least 1 lesion that is measurable using RECIST v1.1 criteria. If the progress is confirmed and meets the RECIST 1.1 standard, it can also be used as target lesion.
6. An expected survival of > 12 weeks.
7. Be able to swallow tablets normally.
8. All acute toxic reactions caused by previous anti-tumor treatment or surgery were relieved to level 0-1 (according to NCI CTCAE version 4.03) or to the level specified in the inclusion / exclusion criteria. Except for other toxicity that researchers think does not pose a safety risk to patients, such as hair loss.
9. Has adequate sufficient organ and bone marrow functions.
10. Fertile female subjects must undergo a serum-negative pregnancy test within 72 hours before starting the study drug and must agree to use a medically approved effective contraceptive during the study period and within 90 days of the last dose of the study drug; Male subjects whose partners are women of child-bearing age should undergo surgical sterilization or agree to use effective methods of contraception during the study period and within 90 days of the last study administration.
11. Patients have agreed and signed the informed consent. Willingness and able to follow the planned visit, research treatment, laboratory examination and other test procedures.

Exclusion Criteria:

1. Known HER2 positive status.
2. The first-line received any taxol drug treatment (if there is tumor recurrence and metastasis during or ≤ 24 weeks after the completion of adjuvant treatment, it is considered that the early-stage adjuvant treatment is a first-line systemic chemotherapy for advanced diseases).
3. Previously received PD-1 / PD-L1 antibody, CTLA-4 antibody, or other small molecular inhibitors for PD-1 / PD-L1 and / or VEGFR.
4. It is known that it is allergic to apatinib, albumin paclitaxel, carrizumab or drug adjuvant; or it has serious allergic reaction to other monoclonal antibodies.
5. Immunosuppressive drugs were used within 14 days before the first use of carrizumab, excluding nasal spray and inhaled corticosteroids or systemic steroids in physiological dose (i.e. no more than 10 mg / day of prednisolone or other corticosteroids in physiological dose of the same drug).
6. The live attenuated vaccine shall be inoculated within 4 weeks before the first administration or during the study period.
7. Central nervous system (CNS) metastasis or presence of brain edema, spinal cord compression, cancerous meningitis, leptomeningeal disease and / or progressive growth. Patients with central nervous system metastases that have been stable for more than 1 month after surgery or radiotherapy can be enrolled in the study if their clinical manifestations are stable 4 weeks after withdrawal of anticonvulsants and steroids before the first administration of the study.
8. The peripheral neuropathy was more than 1 grade.
9. Symptomatic, disseminated to the internal organs, and at risk of life-threatening complications in a short period of time (including patients with uncontrolled large amount of exudate [chest, pericardium, abdominal cavity], lymphangitis and more than 30% of liver involvement).
10. At present, patients with interstitial pneumonia or interstitial lung disease, or with previous history of interstitial pneumonia or interstitial lung disease requiring hormone treatment, or with other pulmonary fibrosis, organic pneumonia (such as bronchiolitis obliterans), pneumoconiosis, drug-related pneumonia, idiopathic pneumonia that may interfere with the judgment and treatment of immune-related pulmonary toxicity, or with active pneumonia on CT at screening stage Patients with severe impairment of pulmonary function; active tuberculosis.
11. There is any active autoimmune disease or a history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or asthma in childhood have been completely relieved, and those who do not need any intervention after adulthood can be included Asthma requiring medical intervention with bronchodilator was not included.)
12. Any other malignant tumor has been diagnosed within 3 years before the study, except for basal cell or squamous cell skin cancer or cervical carcinoma in situ which has been fully treated.
13. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV DNA ≥ 500 IU / ml), hepatitis C (HCV antibody positive, and HCV RNA higher than the detection limit of the analysis method) or co infection with hepatitis B and C.
14. Within 6 months before the study, the following conditions occurred: myocardial infarction, severe / unstable angina, NYHA grade 2 or above cardiac insufficiency, supraventricular or ventricular arrhythmia requiring drug control (including QTc interval > 450 ms for men and 470 MS for women), symptomatic congestive heart failure, cerebrovascular accident (including transient ischemic attack or symptomatic pulmonary embolism).
15. Hypertension, which cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg).
16. Abnormal coagulation (INR > 1.5 or APTT > 1.5 × ULN), bleeding tendency or undergoing thrombolysis or anticoagulation.
17. endencies, such as hemophilia, coagulation skill disorder, thrombocytopenia, hypersplenism and so on.
18. Patients with obvious cough blood or hemoptysis of half teaspoon (2.5ml) or more per day within 2 months before entering the study.
19. In the first 3 months of the study, patients who had significant clinical bleeding symptoms or had definite bleeding tendency, such as gastrointestinal bleeding, bleeding gastric ulcer and positive stool occult blood monitoring twice in the baseline period, should be excluded from gastric bleeding by gastroscope.
20. Events of arteriovenous thrombosis (AVT) occurred within 6 months before the study, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism.
21. Long term anticoagulation with warfarin or heparin or long-term antiplatelet therapy (aspirin ≥ 300 mg / day or clopidogrel > 75 mg / day) is required.
22. Active infection (e.g. intravenous drip of antibiotics, antifungal or antiviral drugs) or fever of unknown origin > 38.5 ° C 2 weeks ago (except for tumor related fever determined by researchers).
23. The history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation is known.
24. Participated in any other drug clinical study within 4 weeks before the first administration, or within 5 half lives from the last study.
25. A history of psychoactive substance abuse or abuse is known.
26. The presence of other serious physical or mental illness or laboratory abnormalities may increase the risk of participating in the study, or interfere with the results of the study, as well as the patients who the investigator believes are not suitable for participating in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity [DLT] | Each 21 days up to Dose-Limiting Toxicity (12-13 months)
  Dose-Limiting Toxicity

SECONDARY OUTCOMES:
Incidence and degree of Adverse Events and Serious Adverse Events [Safety] | Until 30 day safety follow-up visit (Up to 14-18 months)
  Incidence and degree of Adverse Events and Serious Adverse Events
Objective Response Rate [ORR] | Up to 13-16 months
  Objective Response Rate
Duration of response [DoR] | Up to 13-16 months
  Duration of response
Time To Response [TTR] | Up to 13-16 months
  Time To Response
Disease Control Rate [DCR] | Up to13-16 months
  Disease Control Rate
Progression Free Survival [PFS] | Up to 13-16 months
  Progression Free Survival
Overall Survival [OS] | Up to 14-18 months
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: YunPeng Liu, PhD, Principal Investigator — First Hospital of China Medical University
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China

REFERENCES:
- [Result] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Result] Cunningham D, Starling N, Rao S, Iveson T, Nicolson M, Coxon F, Middleton G, Daniel F, Oates J, Norman AR; Upper Gastrointestinal Clinical Studies Group of the National Cancer Research Institute of the United Kingdom. Capecitabine and oxaliplatin for advanced esophagogastric cancer. N Engl J Med. 2008 Jan 3;358(1):36-46. doi: 10.1056/NEJMoa073149. PMID 18172173
- [Result] Catalano V, Graziano F, Santini D, D'Emidio S, Baldelli AM, Rossi D, Vincenzi B, Giordani P, Alessandroni P, Testa E, Tonini G, Catalano G. Second-line chemotherapy for patients with advanced gastric cancer: who may benefit? Br J Cancer. 2008 Nov 4;99(9):1402-7. doi: 10.1038/sj.bjc.6604732. PMID 18971936
- [Result] Li J, Qin S, Xu J, Guo W, Xiong J, Bai Y, Sun G, Yang Y, Wang L, Xu N, Cheng Y, Wang Z, Zheng L, Tao M, Zhu X, Ji D, Liu X, Yu H. Apatinib for chemotherapy-refractory advanced metastatic gastric cancer: results from a randomized, placebo-controlled, parallel-arm, phase II trial. J Clin Oncol. 2013 Sep 10;31(26):3219-25. doi: 10.1200/JCO.2013.48.8585. Epub 2013 Aug 5. PMID 23918952
- [Result] Thuss-Patience PC, Kretzschmar A, Bichev D, Deist T, Hinke A, Breithaupt K, Dogan Y, Gebauer B, Schumacher G, Reichardt P. Survival advantage for irinotecan versus best supportive care as second-line chemotherapy in gastric cancer--a randomised phase III study of the Arbeitsgemeinschaft Internistische Onkologie (AIO). Eur J Cancer. 2011 Oct;47(15):2306-14. doi: 10.1016/j.ejca.2011.06.002. PMID 21742485